CLINICAL TRIAL: NCT02874560
Title: Evaluation of the Functional Remission Occurrence and Predictive Factors in Schizophrenia
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR103490; R092670SCH4033 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: CNS; Antipsychotic; Functional remission; Observational study; FROGS; PSP; Functioning; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Schizophrenia: 350 patients will be included in the study. The centers selection is planned with 100 hospital-based psychiatrists, in centers for preventive medicine (CMP) or in private settings. Each investigator should consecutively enroll patients fulfilling the selection criteria to participate in the study (mean expected number of participants per center is around 10).

SUMMARY:
In a population of patients suffering from schizophrenia being treated for an episode of clinical destabilization and followed for a period of twelve months, the main objective is to evaluate the proportion of patients achieving functional remission and its relationship to clinical remission.

DETAILED DESCRIPTION:
Prospective, national, noninterventional study. One year follow up with three evaluation dates (D0, D180 and D360). The participation of a subject in this study will in no way impact the regular care of the subject or any benefits they are otherwise entitled to. All treatment decisions will be made at the discretion of the participating physician, in accordance with his clinical practice and with approved local prescribing information. Only data available from clinical practice will be collected. Evaluation methods: patient history and clinical examination, clinical global impression (CGI): Improvement in CGI, social performance evaluation [functional remission of general schizophrenia (FROGS scale)], clinical remission evaluation: 8 items of the Positive and negative syndrome (PANSS) Scale, psychosocial remission evaluation (PSP scale), current insight evaluation: insight scale for psychosis, subjective well being under neuroleptic treatment (SWN scale), health condition [Euro quality of life - 5 Dimensions (EQ-5D)]; Judgment Criteria: functional remission is defined as an overall score of greater than or equal to (>=) 57 on the FROGS scale, functional response is defined as improvement of >= 7 points on the FROGS scale. Safety evaluation: no tolerance analysis will be performed, adverse event (AE) and serious adverse event (SAE) with J&J products will be collected and transmitted according to J&J timelines/process.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be male or female adult patients aged 18 to 37 years with a diagnosis of schizophrenia according to diagnostic and statistical manual of mental disorders (DSM-IV) criteria
* Treated for schizophrenia
* Having read understood and signed an informed consent (for patients under legal guardianship, the legal guardian will be informed by the physician)
* Patients must have initiated a long-acting injectable antipsychotic treatment less than 2 months after a previous treatment
* Patients must have been under monitoring by a treatment team from a hospital, a medical psychiatric centre or a clinic for at least 6 months and must be likely to be followed by the same team for the next year

Exclusion Criteria:

* Resistant schizophrenia (no response after receiving two successive antipsychotic treatments at an effective dose, each over at least a four-week period)
* Drug or alcohol dependence or abuse (other than nicotine or caffeine abuse) diagnosed according to DSM-IV in the month preceding the study inclusion process which according to the investigator could compromise the participation in the study
* History of neuroleptic malignant syndrome
* Inability to comply with the requirements of the study (e.g., intellectual deficiency, inability or unwillingness to answer questionnaires) according to the investigator's opinion
* Patients under trusteeship or patient receiving psychiatric care without his consent (except patient under care program)
* Participation in another study within 30 days prior to the study inclusion period

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients are followed in hospital, CMP or clinics for at least 6 months and are likely to be followed by the same team within the next year.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-12 (Actual)

PRIMARY OUTCOMES:
Clinical Remission | 1 year Follow up
  Defined by the absence of a score greater than (>) 3 on the Positive and Negative Syndrome Scale (PANSS) 8 item scale at two consecutive evaluations (D0 and D180 or D180 and D360). The PANSS 8 items allows to evaluate the clinical remission, defined by a score less than or equal to (=<) 3 on each eight items during a six month minimum period. Each of the 8 PANSS items must be scored from 1 (not at all) to 7 (extremely). More the score is high, more the severity rate of the symptom is high.
Functional Remission | 1 year Follow up
  Defined by Functional Remission of General Schizophrenia (FROGS) scale global score and its relationship with clinical remission. FROGS scale: The "Functional Remission of General Schizophrenia" (FROGS) is a 19 items scale gathered in five fields ("Daily life", "Activities", "Adaptation Quality", "relational Life", "Health and treatment") used to evaluate the functional remission in schizophrenia. The 19 items must be scored from 1(not done) to 5 (perfectly done). The total score is 19 to 95. More the score is high, better the functioning abilities are is high.

SECONDARY OUTCOMES:
Functional Response | 1 year Follow up
  Defined as improvement from baseline of greater than or equal to (>=) 7 points on the FROGS scale. FROGS scale: The "Functional Remission of General Schizophrenia" (FROGS) is a 19 items scale gathered in five fields ("Daily life", "Activities", "Adaptation Quality", "relational Life", "Health and treatment") used to evaluate the functional remission in schizophrenia. The 19 items must be scored from 1(not done) to 5 (perfectly done). The total score is 19 to 95. More the score is high, better the functioning abilities are is high.
Satisfactory Level of Functioning | 1 year Follow up
  Defined by the absence of an item less than (<) 3 on the FROGS scale. FROGS scale: The "Functional Remission of General Schizophrenia" (FROGS) is a 19 items scale gathered in five fields ("Daily life", "Activities", "Adaptation Quality", "relational Life", "Health and treatment") used to evaluate the functional remission in schizophrenia. The 19 items must be scored from 1(not done) to 5 (perfectly done). The total score is 19 to 95. More the score is high, better the functioning abilities are is high.
Predictive Clinical Characteristics | 1 year Follow up
  Search for clinical variables predicting an improvement in social performance.
Threshold Score | 1 year Follow up
  Determine a threshold score to define functional remission, satisfactory functioning and optimal functioning on the Mini FROGS scale. Mini FROGS: 4 of the 19 items of FROGS, also scored from 1 (not done) to 5 (perfectly done), the total score is 4 to 20. More the score is high, better the functioning abilities are high.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (1):
- Paris, France